CLINICAL TRIAL: NCT06403358
Title: Prospective Observational Study for the Evaluation of Probiotics Food Supplement in the Re-equilibration of the Intestinal Microbiota, in Paediatric Age
Brief Title: Study for Evaluation of Probiotics in the Re-equilibration of the Intestinal Microbiota, in Paediatric Age
Status: Completed | Type: Observational
Sponsor: Labomar SPA (Industry)
Responsible Party: Sponsor
Other Study IDs: YOV/042022
Record Dates: First submitted 2024-04-19; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: YOVIS BIMBI — 42 male and female subjects, aged between 3 and 14 years with acute diarrhea will be treated with Yovis BAMBINI. The 42 subjects will be recruited with a competitive enrolment at the involved study sites.

SUMMARY:
To evaluate the efficacy, safety and hydration index about the oral administration of probiotics food supplement in the re-equilibration of the intestinal microbiota, in presence of acute diarrhea

DETAILED DESCRIPTION:
Multicenter, observational prospective study evaluating the efficacy, safety and index of hydration resulting from oral administration of probiotics food supplement in paediatric age.

ELIGIBILITY:
Inclusion Criteria:

* • Male and female patients aged between 3 and 14 years;

  * Patients with one of the following conditions:

    * Population with acute diarrhea;
    * Occurrence of at list three liquid or loose stools per day;
    * Consistency of stools (≥ type 5) according to Bristol Stool Scale Form (BFS).
  * Informed consent signed by parents or the patient's legal guardian(s) for study enrollment.

Exclusion Criteria:

* • Presence of chronic diarrhea characterized by the emission of poorly formed stools, for more than 4 weeks, accompanied by increased frequency of evacuation or urgency to defecation;

  * Known or potential hypersensitivity and/or history of allergic reactions to one of the components of probiotics food supplement;
  * Coexisting severe infection (e.g. sepsis, pneumonia, meningitis);
  * Patients affected by chronic intestinal disease, immune deficiency, neurological disease and tumors;
  * Contemporary consumption of other probiotics compounds;
  * Patients whose parents or the patient's legal guardian(s)refuse to provide written informed consent;
  * Patient who has not expressed his consent according to his age and level of understanding;
  * Participation in another clinical trial within the previous 30 days;
  * Evidence of severe or uncontrolled systemic disease or any other significant disorders, which in the opinion of the investigator does not allow the participation in the study or could compromise the results

Ages: 3 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: 42 male and female subjects, aged between 3 and 14 years with acute diarrhea will be treated with Yovis BAMBINI. The 42 subjects will be recruited with a competitive enrolment at the involved study sites.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of oral administration of probiotics food supplement in paediatric population with acute diarrhea | Baseline, during the intervention, immediately after the intervention
  Reduction of the number of loose stools per day
Evaluation of the efficacy of oral administration of probiotics food supplement in paediatric population with acute diarrhea | Baseline, during the intervention, immediately after the intervention
  Reduction of diarrhea duration.

SECONDARY OUTCOMES:
Evaluation of the safety profile of probiotics food supplement | Immediately after the intervention
  Investigator Global Assessment of Safety (IGAS): using the 4-point scale:1= very good safety, 2 =good safety, 3 = moderate safety and 4 = poor safety. IGAS will be evaluated at the last visit.
Evaluation of the safety profile of probiotics food supplement | During the intervention, immediately after the intervention
  Evaluation of the eventual presence adverse event/serious adverse events.
Assessment of the compliance to the treatment | During the intervention, immediately after the intervention
  Compilation of the daily diary to the family;Compilation of the degree satisfaction questionnaires to the family;Compilation of the degree satisfaction questionnaires to the patient
Analysis of the hydration state | BaselinaDuring the intervention, immediately after the intervention
  Degree of dehydration using the Gorelick scale: using the 10-point score: 0 to 3 (mild dehydration), 3 to 5 (moderate dehydration), 6 to 10 (severe dehydration); Change in body weight;

CONTACTS AND LOCATIONS:
Locations (1):
- Studio Pediatrico Dr. Gaetano Bottaro, Gravina di Catania, Catania, Italy